CLINICAL TRIAL: NCT01957995
Title: An Open Label, Randomized Study to Evaluate Safety and Pharmacokinetics of Intravenous Infusion of Nanosomal Docetaxel Lipid Suspension for Injection in Patients With Advanced Solid Tumors
Brief Title: Nanosomal Docetaxel Lipid Suspension in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Jina Pharmaceuticals Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0C-13-2; NCI-2013-01731 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 022-13; 0C-13-2 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (lowest dose NDLS) (Experimental): Patients receive lowest dose nanosomal docetaxel lipid suspension IV over 1 hour.
  Interventions: Drug: nanosomal docetaxel lipid suspension; Other: pharmacological study
- Arm II (low dose NDLS) (Experimental): Patients receive low dose nanosomal docetaxel lipid suspension IV over 1 hour.
  Interventions: Drug: nanosomal docetaxel lipid suspension; Other: pharmacological study
- Arm III (high dose NDLS) (Experimental): Patients receive high dose nanosomal docetaxel lipid suspension IV over 1 hour.
  Interventions: Drug: nanosomal docetaxel lipid suspension; Other: pharmacological study
- Arm IV (highest dose NDLS) (Experimental): Patients receive highest dose nanosomal docetaxel lipid suspension IV over 1 hour.
  Interventions: Drug: nanosomal docetaxel lipid suspension; Other: pharmacological study

INTERVENTIONS:
Drug: nanosomal docetaxel lipid suspension — Given IV
Other: pharmacological study — Correlative studies

SUMMARY:
This randomized phase I trial studies the side effects and best dose of nanosomal docetaxel lipid suspension in treating patients with advanced solid tumors. Drugs used in chemotherapy, such as nanosomal docetaxel lipid suspension, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the pharmacokinetics profile of nanosomal docetaxel lipid suspension (NDLS) in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To assess the safety and toxicity of NDLS in patients with advanced solid tumors.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive lowest dose nanosomal docetaxel lipid suspension intravenously (IV) over 1 hour.

ARM II: Patients receive low dose nanosomal docetaxel lipid suspension IV over 1 hour.

ARM III: Patients receive high dose nanosomal docetaxel lipid suspension IV over 1 hour.

ARM IV: Patients receive highest dose nanosomal docetaxel lipid suspension IV over 1 hour. In all arms, treatment may repeat every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written, personally signed and dated, informed consent to participate in the study before initiating any study related procedures
* Body mass index (BMI) at least 17 calculated as weight in kg/height in m^2
* Must have histopathologically/cytologically confirmed primary tumors for which docetaxel is an appropriate or reasonable treatment option
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Must have recovered from any toxic effects of previous chemotherapy or radiotherapy as judged by the investigator to =< grade 1
* Previous chemotherapy/radiotherapy/targeted therapy should have been completed at least 4 weeks prior to start of NDLS administration
* Life expectancy of at least 6 months
* Female patients of child bearing potential must have negative serum pregnancy test at screening
* Sexually active women, unless surgically sterile (at least 6 months prior to study drug administration) or postmenopausal for at least 12 consecutive months, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to study drug administration] sexual partner) for at least 4 weeks prior to study drug administration, during study and up to 30 days after the last dose of study drug; cessation of birth control after this point should be discussed with a responsible physician
* In case of male patients: either patient partners or patients themselves must use an effective method of avoiding pregnancy for at least 4 weeks prior to study drug administration, during study and up to 30 days after the last dose of study drug or till next chemotherapy cycle
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9 gm/dl
* Serum creatinine < 1.5 times upper limit of normal (ULN)
* Total bilirubin =< ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5X ULN if alkaline phosphatase < 2.5 ULN
* AST/ALT < 1.5 X ULN if alkaline phosphatase > 2.5 ULN
* Alkaline phosphatase must be < 5 x ULN on all cases

Exclusion Criteria:

* Hypersensitivity to docetaxel injection or any of its excipients
* Intolerance to any antineoplastic agents belonging to the taxane family
* Prior anticancer therapy within 28 days prior to the first day of study treatment
* Participation in another experimental drug study within 30 days prior signing the informed consent form (ICF)
* Any of the following cardiac conditions:

  * Unstable angina
  * Myocardial infarction within the past 6 months
  * New York State Heart Association (NYHA) class II-IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Clinically significant pericardial disease
  * Electrocardiographic evidence of acute ischemic or active conduction system abnormalities
  * Evidence of abnormal cardiac conduction (e.g., bundle branch block or heart block) are eligible if their disease has been stable for the past six months * History of cardiac disease that met the NYHA classification class 2 or greater
* Use of any recreational drugs or history of drug addiction
* Known history of brain metastasis
* Pre-existing motor or sensory neurotoxicity of a severity >= grade 2 by National Cancer Institute (NCI) criteria
* Positive hepatitis screening (hepatitis screen includes hepatitis B surface antigen [HBsAg], hepatitis C virus [HCV] and hepatitis A virus [HAV] [immunoglobulin M (IgM)] antibody)
* Known case of active infection including human immunodeficiency virus (HIV) infections
* Any other condition that, in the investigator's judgment, might increase the risk to the patient or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study
* Abnormal baseline findings considered by the investigator to indicate conditions that might affect study endpoints
* Donation of blood (1 unit or 350 mL) within 90 days prior to receiving the first dose of study medicine
* Known, existing uncontrolled coagulopathy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2014-05-29 (Actual); Study Completion 2016-07-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of nanosomal docetaxel lipid suspension | Pre-dose and post dose at 10, 20, 30, 40, 50, 60, 80, and 100 minutes and 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, and 48 hours
  Descriptive statistics of all pharmacokinetic parameters would be computed and reported for free and total docetaxel. Maximum blood concentration (Cmax), area under the curve (AUC)0-t, AUC0-infinity, time to Cmax (Tmax), terminal elimination rate constant (lambda z), half-life (t1/2), AUC percent extrapolated (%Extrap), clearance (CL), and volume of distribution (Vd) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States